CLINICAL TRIAL: NCT01676272
Title: Proposal for a Multi- Center Site Randomized, Prospective Controlled Head-to-head Clinical Trial Comparing a Bioengineered Skin Substitute to a Human Skin Allograf
Brief Title: Multi Center Site , Controlled Trial Comparing a Bioengineered Skin Substitute to a Human Skin Allograft
Status: Completed | Type: Observational
Sponsor: Solsys Medical LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: soluble 102
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2015-11

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Despite the widespread use of advanced biologics for the treatment of diabetic foot ulcers, data comparing one type of modality to another are scarce. This investigation is a prospective randomized study comparing a bioengineered skin substitute to a human skin allograft.

DETAILED DESCRIPTION:
The primary goal in treating a DFU is to obtain wound closure. Healing can be a lengthy and painful process for ulcers of diabetic etiology. Healing is often further complicated in subjects with diabetes by vascular compromise and peripheral ischemia, renal insufficiency and diminution of inflammatory responses

The two products to be compared in this study are both commonly used for the treatment of diabetic foot ulcers. DermaGraft is considered a medical device by the FDA, and was cleared for the treatment of diabetic foot ulcers in 1997. It is a staple for the treatment of diabetic foot ulcers, and is widely used throughout the United States. It is composed of an absorbable substrate that has been seeded with living human fibroblasts. Once formed, the graft is cryopreserved until it reaches the clinic, where it is defrosted and applied to the wound surface.

TheraSkin is composed of a split thickness skin graft harvested within 24 hours post-mortem, from an organ donor who has cleared the standard safety screenings. It is classified by the FDA as a donated tissue. Once harvested, the graft is sanitized according to FDA specifications, and cryopreserved, until it is delivered to the clinic for application to the foot ulcer. It is also a widely used treatment for diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:: Subjects are required to meet all of the following criteria for enrollment into the study and subsequent randomization.

1. A signed and dated informed consent form has been obtained from the subject.
2. Subject is able and willing to comply with study procedures
3. Subject is male or female and is 18 years of age or older.
4. Subject, if female of childbearing potential, has a negative serum pregnancy test at screening
5. Subject has type 1 or type 2 diabetes mellitus
6. Subject has glycosylated hemoglobin, HbA1c, less than or equal to 12%
7. Presence of at least one DFU that meets all of the following criteria:

   1. Ulcer has been diagnosed as a full-thickness DFU and including those of the heel.
   2. There is a minimum 2 cm margin between the qualifying study ulcer and any other ulcers on the specified foot, post-debridement)
   3. Ulcer size (area) greater than 1 cm2 (post-debridement at time of randomization) not deeper than 5mm. deep. Ulcer size no larger than 10 cm2
   4. Wagner grade 1 at initialization of the clinical trial
   5. Duration of the study ulcer is at least 30 days at the time of the screening visit Note: If the subject has more than one qualifying DFU, the ulcer designated as the study ulcer will be at the discretion of the Investigator.
8. Subject has adequate vascular perfusion of the affected limb, as defined by at least one of the following:

   1. Ankle-Brachial Index (ABI) at least 0.65 (moderate arterial disease) and less than1.2
   2. Toe pressure (plethysmography) > 50 mm Hg
   3. TcPO2 > 40 mm Hg
   4. Doppler ultrasound (biphasic or triphasic waveforms) consistent with adequate bloodflow to the affected extremity, as determined by the Investigator
9. Standard of Care practices of the Investigator and the site:

Subject or responsible caregiver is willing and able to maintain the required off-loading (as applicable for the location of the ulcer) and applicable dressing changes.

-

Exclusion Criteria:Subjects meeting any of the following criteria will be excluded from enrollment and subsequent randomization.

1. Subject has suspected or confirmed signs/symptoms of gangrene or wound infection on any part of the affected limb. (Subjects with wound infection at the screening visit may be treated and re-screened for participation in the study after eradication of the infection).
2. Subject has a history of hypersensitivity to bovine collagen and/or chondroitin, as listed in the Dermagraft Directions for Use.
3. Subject has a history of hypersensitivity to any of the antibiotics or preservation agents listed in the TheraSkin Instructions for Use.
4. Subject cannot be pregnant at the time of treatment.
5. Subject was previously treated under this clinical study protocol.
6. Subject has participated in another clinical trial involving a device or a systemically administered investigational study drug/treatment within 30 days of randomization visit.
7. Subject is currently receiving (i.e., within 30 days of randomization visit) or scheduled to receive a medication or treatment which, in the opinion of the Investigator, is known to interfere with or affect the rate and quality of wound healing (e.g., systemic steroids, immunosuppressive therapy, autoimmune disease therapy, cytostatic therapy within the 12 months prior to randomization, dialysis, radiation therapy to the foot, vascular surgery, angioplasty or thrombolysis).
8. Subject has any of the following unstable conditions or circumstances that could interfere with treatment regimen compliance:

   1. Ability to perform required dressing changes
   2. Ability to comply with treatment visit schedule
   3. Mental incapacity
   4. Current substance abuse
9. Subject has excessive lymphedema, which, in the opinion of the Investigator, could interfere with wound healing.
10. Subject has unstable Charcot foot or Charcot with boney prominence that, in the opinion of the Investigator, could inhibit wound healing.
11. Subject has ulcers secondary to a disease other than diabetes, e.g., vasculitis, neoplasm's, or hematological disorders.
12. Subject has osteomyelitis with necrotic soft bone. (If the Investigator suspects the presence of osteomyelitis, the diagnosis must be confirmed by plain film X-ray.)
13. Subject with Chopart amputation.
14. Subject has a history of bone cancer or metastatic disease on the affected limb, radiation therapy to the foot or has had chemotherapy within the 12 months prior to randomization.
15. Subject has been treated with wound dressings that include growth factors, engineered tissues, or skin substitutes (e.g., Regranex®, Dermagraft®, Apligraf®,Theraskin® GraftJacket®, OASIS®, Primatrix®, Matristem®,etc.) within 30 days of randomization.
16. Subject has been treated with hyperbaric oxygen within 5 days of screening.
17. Subject has a history of or any of the following current illnesses or conditions (other than diabetes) that would compromise the safety of the subject, or the normal wound healing process:

    1. End-stage renal disease
    2. Immunosuppression
    3. Severe malnutrition
    4. Liver disease
    5. Aplastic anemia
    6. Scleroderma
    7. Acquired immune deficiency syndrome (AIDS) or HIV positive
    8. Connective tissue disorder
    9. Exacerbation of sickle cell anemia
18. Subject is an employee or relative of any member of the Investigational site or the Sponsor.

    -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes Diabetic patients with type 1 or type 2 Diabetes with foot ulcers
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2012-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Proposal for a multi center site randomized, prospective controlled head-to-head clinical trial comparing a bioengineered skin substitute to a human skin allograft. | 2 years
  Despite the widespread use of advanced biologics for the treatment of diabetic foot ulcers, data comparing one type of modality to another are scarce. This investigation is a prospective randomized study comparing a bioengineered skin substitute to a human skin allograft.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Keller, DPM, Principal Investigator — Mary Immaculate Hospital
Locations (2):
- United States (2):
  - Washington Hospital Wound Center, Washington, Pennsylvania
  - Mary Immaculat Hospital Wound Care Center, Newport News, Virginia